CLINICAL TRIAL: NCT06559280
Title: The Effect of Subclinical Doses of Ketamine on Early Postoperative Pain Sensitivity in Patients Undergoing Salpingectomy: a Prospective, Double-blind, Randomized Controlled Clinical Trial
Brief Title: The Effect of Subclinical Dose of Ketamine on Early Postoperative Pain Sensitivity in Patients Undergoing Salpingectomy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Wu Yanqin, physician, Fujian Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: K2023-11-022
Record Dates: First submitted 2024-08-11; First posted 2024-08-19 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Ectopic Pregnancy
MeSH Terms: conditions — Pregnancy, Ectopic | interventions — Esketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Use ketamine for postoperative analgesia and intraoperative induction
  Interventions: Drug: esketamine
- control group (No Intervention): Not using ketamine for postoperative analgesia and intraoperative induction

INTERVENTIONS:
Drug: esketamine — During the operation, 0.25mg/kg esketamine was induced, and 1mg/kg esketamine was added to the postoperative analgesia pump
  Arms: experimental group

SUMMARY:
The experiment aims to explore the clinical effect of subclinical doses of ketamine on early postoperative pain sensitivity in ectopic pregnancy population.

DETAILED DESCRIPTION:
Ectopic pregnancy (EP) refers to the implantation and development of a fertilized egg outside the uterine cavity, and is one of the common acute abdominal conditions in obstetrics and gynecology. Among them, tubal pregnancy is the most common type, with the highest incidence rate among all ectopic pregnancies. After falling ill, it is easy for patients to experience symptoms such as vaginal bleeding, abdominal pain, and amenorrhea, and even infertility, which seriously affects their physical and mental health. After diagnosis, patients often experience negative emotions such as anxiety, fear, and depression. A history of preoperative anxiety and depression can lower the patient's pain threshold, leading to poor postoperative pain control. In gynecological laparoscopic surgery, ectopic pregnancy surgery is also a relatively painful type of surgery, and the establishment of pneumoperitoneum during surgery can easily cause postoperative pain and affect the patient's prognosis and quality of life. And the patient's preoperative preparation time is limited, leading to a decrease in pain tolerance and an increased demand for postoperative analgesia . Therefore, the issue of increased postoperative pain sensitivity in patients with ectopic pregnancy deserves attention.

Ketamine is an N-methyl-D-aspartate (NMDA) receptor inhibitor that can effectively inhibit NMDA receptor-mediated central sensitization. As an adjuvant analgesic for preventing postoperative hyperalgesia induced by remifentanil, it has a definite therapeutic effect . Esketamine, also known as right ketamine, has pharmacological characteristics similar to racemic ketamine while enhancing analgesic and sedative effects, helping to reduce perioperative opioid use. It has also shown significant advantages in the treatment of pain sensitivity, depression, and epilepsy . However, there are relatively few studies on the postoperative pain sensitivity of subclinical doses of ketamine and ectopic pregnancy patients in clinical practice, and whether it can improve postoperative pain sensitivity in such patients still needs further research and exploration.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years old
* BMI 18-30 kg/m2;
* American Society of Anesthesiologists (ASA) classification I and II
* The patient was diagnosed with ectopic pregnancy through ultrasound examination, and it was confirmed that there was no embryo or gestational sac in the uterus; The patient has indications for laparoscopic ectopic pregnancy surgery;
* All patients are scheduled to undergo laparoscopic salpingectomy for treatment Normal mental state;
* No cognitive impairment;
* Normal communication skills, no speech barriers

Exclusion Criteria:

* Individuals with severe organ dysfunction such as heart, lungs, liver, and kidneys;
* Individuals with serious mental illnesses;
* Long term use of sedatives and analgesics or long-term alcoholism and smoking;
* History of allergy to ketamine and related drugs
* There is a serious risk of hypertension or elevated intracranial pressure, as well as contraindications for the use of ketamine in cases of hyperthyroidism Refuse to join the trial;
* Patients with a history of other chronic pain diseases.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-08-24 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Postoperative pain sensitivity | Preoperative, one day after surgery, the second day after surgery, and one week after surgery
  The pain sensitivity scale is used to measure the pain sensitivity of patients. Patients imagine certain scenarios in their daily lives and score their pain to evaluate their individual pain sensitivity. This scale contains 17 items, requiring testers to fill in a number on the numerical rating scale from 0 (no pain) to 10 (most pain) to indicate the degree of pain in this situation. There are three items interspersed among them that describe situations where there is no pain under normal circumstances, as a reference for testers to feel no pain. In addition, the 14 pain items cover various types of pain and pain intensity levels, and completing the PSQ generally takes 5-10 minutes. The total score of PSQ is based on the average score of 14 pain items, ranging from 0 to 10. The results are divided into two categories: PSQ moderate and PSQ minor, which reflect the expected pain levels of different intensity stimuli. The higher the score, the more sensitive it is to pain stimuli.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuzhou University affiliated Provincial Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No